CLINICAL TRIAL: NCT05004220
Title: Studie Vlivu darování krevní Plazmy - Plasmapheresis. Study of the Plasma Donation Effect - Plasmapheresis
Brief Title: Effects of Plasmapheresis on Aging Biomarkers
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Hradec Kralove (Other); Longevitytech.fund a.s. (Unknown); Clock Foundation (Unknown); AGECURVE LIMITED (Unknown)
Responsible Party: Principal Investigator, Pavel Borsky, M.D., Charles University, Czech Republic
Other Study IDs: 202103 P07
Record Dates: First submitted 2021-07-30; First posted 2021-08-13 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Aging; Plasmapheresis
Keywords: Aging; Plasmapeheresis
MeSH Terms: interventions — Plasmapheresis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 consists of first time donors undergoing all 8 tracked plasmaphereses.
  Interventions: Procedure: Plasmapheresis
- Group 2: Group 2 consists of first time donors undergoing only last 4 plasmaphereses, serving as control for the first 4 donations.
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Procedure: Plasmapheresis — Procedure whereby plasma is separated and extracted from anticoagulated whole blood and the red cells retransfused to the donor.

SUMMARY:
The aim of the study is to evaluate the effect of plasmapheresis (repeated plasma withdrawals) on selected health indicators (hematological, biochemical, immunological and indicators of biological age) of plasma donors.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy volunteer subjects age 40 - 60
2. 50:50 man and woman

Exclusion Criteria:

1. Subjects excluded from plasma donation protocols (serious illness, infection, etc)
2. Subjects undergoing stronger anti-aging interventions

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 41 donors are welcomed to begin with the study. The participants are divided into 2 groups (Group 1 = therapeutic, Group 2 = half control) using stratified randomization, major criteria being chronological age and BMI, minor criteria being illness/medication, smoking, COVID in past 3 months, covid vaccination.
  Group 1 consists of 28 participants (14 female, 14 male). Group 2 consists of 13 participants (7 female, 6 male). We suppose that the number of participants will decline during each phase of the study, approx. 10% before it even starts, 10% in the middle, 10% in the end. The goal is to have more than 30 participants finishing the study.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Significant change of biological age according to epigenetic clock after 8 plasmaphereses | Through study completion, an average of 8 months
  Significant change of the epigenetic age of the plasma donors after 8 cycles of plasmapheresis conducted or a slower increase of the biological age throughout the study than the increase of the chronological age.

SECONDARY OUTCOMES:
Significant change of biological age according to epigenetic clock after 8 plasmaphereses | Through study completion, an average of 8 months
  Significant change of the epigenetic age of the plasma donors after 4 cycles of plasmapheresis conducted or a slower increase of the biological age throughout the study than the increase of the chronological age.
Significant change of the proteomic profile after 8 plasmaphereses | Through study completion, an average of 8 months
  Proteomic analysis showing signs of a rejuvenated proteostasis in the plasma donors after 8 cycles of plasmapheresis.
Significant change of the proteomic profile after 4 plasmaphereses | Through study completion, an average of 8 months
  Proteomic analysis showing signs of a rejuvenated proteostasis in the plasma donors after 8 cycles of plasmapheresis.
Significant change of the biological age according to a blood biochemistry clock after 8 plasmaphereses | Through study completion, an average of 8 months
  Blood biochemistry clock showing phenotype of a younger individual in the plasma donors after 8 cycles of plasmapheresis.
Significant change of the biological age according to a blood biochemistry clock after 4 plasmaphereses | Through study completion, an average of 8 months
  Blood biochemistry clock showing phenotype of a younger individual in the plasma donors after 8 cycles of plasmapheresis.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles University, Medical Faculty in Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No